CLINICAL TRIAL: NCT07236086
Title: Evaluating the Analgesic Efficacy of Superficial Cervical Plexus Block for Maxillofacial Surgeries : A Comparative Randomized Control Study
Brief Title: Evaluating the Analgesic Efficacy of Superficial Cervical Plexus Block for Maxillofacial Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rahma Mohamed Atef Mohamed, Principle Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCPB267
Record Dates: First submitted 2025-09-28; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Maxillofacial Surgeries
MeSH Terms: interventions — small cardioactive peptide B; Sodium Chloride; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient, surgeon, the outcome assessor and the statistician will be blinded about patient's group allocation. The anesthetist responsible for the patient intraoperatively will not be blinded to patient group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): patients will recive IV saline only
  Interventions: Drug: Saline (0.9% NaCl)
- study group (Active Comparator): patient will recived superficial Cervical plexus Block with 10 mL of 0.25% bupivacaine
  Interventions: Procedure: superficial cervical plexus nerve block; Drug: Bupivacaine

INTERVENTIONS:
Procedure: superficial cervical plexus nerve block — The fascial plane delineating the space between the levator scapulae and SCM can then be detected. Within this striated, hyperechoic substance, a hypoechoic cluster representing the superficial cervical plexus can be visualized, typically located just deep to the posterior surface of the lateral SCM.
  With an in-plane technique, 22-G needle is introduced parallel to the ultrasound beam, proceeding from the posterolateral to the medial direction. The needle will be advanced through the skin and platysma under real-time ultrasound guidance until it approaches to the plexus. Aspiration will be performed to ensure the needle tip is not within a vascular structure.
  Other Names: SCPB
  Arms: study group
Drug: Saline (0.9% NaCl) — patient will recive saline
  Arms: control group
Drug: Bupivacaine — 10 mL of 0.25% bupivacaine will be administered in a supine position with the head turned opposite to the side of the block.
  Arms: study group

SUMMARY:
The superficial cervical plexus (SCP) originates from the anterior rami of C1-C4 and gives four cutaneous branches supplying the anterolateral neck, external ear, and shoulder tip (1). A superficial cervical plexus block (SCPB) is performed by subcutaneous injection at the midpoint of the posterior border of the sternocleidomastoid, targeting these sensory branches using either landmarks or ultrasound guidance. The goal of the ultrasound (US)-guided technique of superficial cervical plexus nerve block is to deposit local anesthetic within the vicinity of the sensory branches of the nerve roots C2, C3, and C4 (2). SCPB has been successfully used for analgesia in mandibular, tympanomastoid, thyroid, submandibular, and clavicular surgeries, and can even serve as the sole anaesthetic technique in external ear procedures (3, 4). As complications may arise while administrating a SCPB, an adequate understanding of the block physiology and local anesthetic toxicity can mitigate these issues. Superficial cervical plexus block shares common complications with other local anesthetic-based nerve blocks including intravascular injection into a vein or an artery, hematoma formation, infection risk and local anesthetic toxicity. It is worthy to refer that complications are of a higher incidence in deep blocks than superficial ones

DETAILED DESCRIPTION:
The superficial cervical plexus (SCP) originates from the anterior rami of C1-C4 and gives four cutaneous branches supplying the anterolateral neck, external ear, and shoulder tip (1). A superficial cervical plexus block (SCPB) is performed by subcutaneous injection at the midpoint of the posterior border of the sternocleidomastoid, targeting these sensory branches using either landmarks or ultrasound guidance. The goal of the ultrasound (US)-guided technique of superficial cervical plexus nerve block is to deposit local anesthetic within the vicinity of the sensory branches of the nerve roots C2, C3, and C4 (2). SCPB has been successfully used for analgesia in mandibular, tympanomastoid, thyroid, submandibular, and clavicular surgeries, and can even serve as the sole anaesthetic technique in external ear procedures (3, 4). As complications may arise while administrating a SCPB, an adequate understanding of the block physiology and local anesthetic toxicity can mitigate these issues. Superficial cervical plexus block shares common complications with other local anesthetic-based nerve blocks including intravascular injection into a vein or an artery, hematoma formation, infection risk and local anesthetic toxicity. It is worthy to refer that complications are of a higher incidence in deep blocks than superficial ones .

Based on this background, the present study aims to evaluate the analgesic effect of US-guided SCPB in maxillofacial surgeries compared with conventional general anaesthesia, focusing on intra- and postoperative systemic analgesic requirements, pain scores on the visual analog scale (VAS), total duration of analgesia, vital parameters, and the incidence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18-65 years

  * BMI < 30 kg/m2
  * American Society of Anesthesiologists physical status classification (ASA) I - III
  * Patients scheduled for maxillofacial procedures involving submandibular area e.g. submandibular and submental abscesses, neck region e.g. cervical lymph node biopsies and ear lobe procedures.

Exclusion Criteria:

* • Patient refusal

  * Coagulopathy
  * Local infection ate the site of injection
  * Pre-existing neuropathy or neurological disease
  * Hypersensitivity to local anaesthetics used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
the first call for rescue analgesia | 24 HOURS
  the elapsed time from the time of block until the first postoperative analgesic use after the end of the surgery, which will be administrated based on patient request

SECONDARY OUTCOMES:
The total analgesic requirement | 24 hours.
  The total analgesic requirement of Nalbuphine in mg given postoperatively
Pain scores; Visual Analouge Scale (VAS) score | 24 hours
  visual analogue scale (VAS) at rest and when coughing postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Rahma M. Atef, MBBCH, Principal Investigator — Assiut University